CLINICAL TRIAL: NCT03691766
Title: Effect of Photobiomodulation Therapy on Muscle Function and Inflammation in Persons With Multiple Sclerosis
Brief Title: Photobiomodulation Therapy in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: University of Wisconsin, Milwaukee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HR-1710020115
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation Therapy (Experimental): Experimental: Photobiomodulation Therapy comprising 640 nm, 875 nm, and 905 nm light (red lights)
  Interventions: Other: Photobiomodulation Therapy
- Control (Placebo Comparator): Placebo device with different wavelengths of light without known physiologic effect.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Photobiomodulation Therapy — Photobiomodulation therapy, a mix of red lights thought to improve mitochondrial function will be applied in and acute and chronic manner to test whether muscle fatigue improves in persons with MS.
  Arms: Photobiomodulation Therapy
Other: Placebo — Device with sham light source
  Arms: Control

SUMMARY:
This study will test whether photobiomodulation therapy improves muscle endurance and decreases inflammation in persons with relapsing-remitting multiple sclerosis. We will also investigate mechanisms for any improvements.

DETAILED DESCRIPTION:
Persons with multiple sclerosis (MS) MS commonly experience muscle weakness and fatigue which may contribute to the commonly reported symptomatic fatigue. Photobiomodulation therapy (PBMT) induced with light in the visible red to near infrared (VIS/NIR) region of the spectrum (600-1000 nm) can stimulate cytochrome c oxidase and improve mitochondrial function. PBMT is an emerging therapeutic modality for soft tissue injury, chronic inflammation, neurodegeneration , and retinal diseases. PBMT has also been used to enhance muscle endurance, strength and recovery in healthy adults. We propose that in persons with MS, PBMT will 1) enhance regional muscle endurance after acute treatment and 2) enhance functional endurance after extended treatment. We will also test to determine if improvements are due to central or peripheral neuromuscular or cardiovascular mechanisms. Final, we will explore if regional PBMT can result in systemic anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsing remitting MS,
2. Independent or ambulatory with minimal aid.
3. Must be able to move foot (ankle dorsiflexion) at least moderately forcibly against gravity (manual muscle test score 3-5)
4. Subjects must be able to walk for 6 minutes independently with no or minimal use of an assistive device.

Exclusion Criteria:

1. No noticeable left right ankle strength asymmetry
2. No exacerbations (MS attacks) or immunosuppressive therapy use within the previous 6 months
3. No concurrent infection or known cardiovascular disease including having a pacemaker; or other serious medical co-morbidity including metabolic, mitochondrial, autoimmune, diseases or other co-existing neurologic conditions.
4. Not involved in any clinical trial or other research that could confound results.
5. Must not be pregnant
6. Must not have an active diagnosis of cancer

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Muscle Fatigue | up to 4 week photobiomodulation intervention, immediately after the intervention, and then 4 months after this extended treatment
  Change in muscle fatigue or recovery after photobiomodulation therapy

SECONDARY OUTCOMES:
Systemic Inflammation | up to 4 week photobiomodulation intervention, and then again at 4 months post-intervention
  Change in pro- and anti-inflammatory cytokines.

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No